CLINICAL TRIAL: NCT02129595
Title: Effects of Resveratrol on Insulin Sensitivity, Brown Adipose Tissue and Metabolic Profile in First-degree Relatives of Type 2 Diabetic Patients
Brief Title: Resveratrol and First-degree Relatives of Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry); Diabetes Fonds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13-3-058
Record Dates: First submitted 2014-04-24; First posted 2014-05-02 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2016-08

CONDITIONS: Pre-diabetes
Keywords: Resveratrol; Diabetes Mellitus; Diabetes Mellitus, Type 2; Insulin Resistance; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Hyperinsulinism; Anti-Inflammatory Agents, Non-Steroidal; Analgesics, Non-Narcotic; Analgesics; Sensory System Agents; Peripheral Nervous System Agents; Physiological Effects of Drugs; Pharmacologic Actions; Anti-Inflammatory Agents; Therapeutic Uses; Antirheumatic Agents; Antineoplastic Agents, Phytogenic; Antineoplastic Agents; Antioxidants; Molecular Mechanisms of Pharmacological Action; Protective Agents; Enzyme Inhibitors; Platelet Aggregation Inhibitors; Hematologic Agents; Antimutagenic Agents; Anticarcinogenic Agents; Central Nervous System Agents; Brown Adipose Tissue
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus; Diabetes Mellitus, Type 2; Insulin Resistance; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Hyperinsulinism | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- resveratrol (Active Comparator): resveratrol will be given for 30 or 34 days (if included in brown adipose tissue measurement), twice daily. One pill, which contains 75 mg of resveratrol, will be provided with lunch, and the other pill of 75 mg will be provided with dinner. So in total 150 mg/day of resveratrol will be given.
  Interventions: Dietary Supplement: resveratrol
- placebo (Placebo Comparator): A placebo will be given for 30 or 34 days (if included in brown adipose tissue measurement), twice daily. One pill will be provided with lunch and the other pill will be provided with dinner.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: placebo — A placebo will given for 30 days or 34 days (if included in brown adipose tissue measurement), twice daily. One pill will be provided with lunch, and the other pill will be provided with dinner.
  Arms: placebo
Dietary Supplement: resveratrol — resveratrol will be given for 30 days or 34 days (if included in brown adipose tissue measurement), twice daily. One pill, which contains 75 mg of resveratrol, will be provided with lunch, and the other pill, also containing 75 mg will be given with dinner. So in total a dose of 150 mg/day will be given.
  Other Names: resVida (99% pure trans-resveratrol)
  Arms: resveratrol

SUMMARY:
The main objective of the study is to investigate if resveratrol supplementation can improve overall and muscle-specific insulin sensitivity in first-degree relatives of type 2 diabetic patients.

As a secondary objective the investigators want to investigate whether the improved insulin sensitivity can be attributed to improved muscle mitochondrial oxidative capacity and a reduced intrahepatic and cardiac lipid content. Furthermore, in a subset of the participants the investigators want to investigate the effect of resveratrol on glucose uptake in brown adipose tissue.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age: 40-70 years
* BMI 27-35 kg/m2
* Has first-degree relative(s) diagnosed with type 2 diabetes
* Sedentary
* Not more than 2 hours of sports a week
* No active job that requires strenuous physical activity
* Stable dietary habits: no weight gain or loss > 5kg in the last three months
* Insulin resistant: glucose clearance rate below < 350 ml/kg/min, as determined using OGIS120
* Willingness to abstain from resveratrol-containing food products
* Subjects will only be included when the dependent medical doctor of this study approves participation after evaluating data obtained during screening

Exclusion Criteria:

* Use of anticoagulants
* Uncontrolled hypertension
* Haemoglobin <7.8 mmol/l
* In case of an abnormal ECG in rest: this will be discussed with the responsible medical doctor
* HBA1C > 6.5%
* Diagnosed with type 2 diabetes
* Medication use known to interfere with glucose homeostasis/metabolism
* Current alcohol consumption > 20 grams/day
* Subjects who don't want to be informed about unexpected medical findings during the screening /study, or do not wish that their physician is informed, cannot participate in the study.
* Subjects who intend to donate blood during the intervention or subjects who have donated blood less than three months before the start of the intervention.
* Participation in another biomedical study within 1 month before the first screening visit
* Any condition, disease or abnormal laboratory test result that, in the opinion of the Investigator, would interfere with the study outcome, affect trial participation or put the subject at undue risk
* Any contra-indication to MRI scanning. These contra-indications include patients with following devices:

  * Central nervous system aneurysm clip
  * Implanted neural stimulator
  * Implanted cardiac pacemaker of defibrillator
  * Cochlear implant
  * Insulin pump
  * Metal containing corpora aliena in the eye or brains

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04; Primary Completion 2017-04 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity: overall, muscle- and liver specific | 30 days after supplementation
  Hyperinsulinemic euglycemic clamp combined with indirect calorimetry: Glucose infusion rate (GIR), rate of appearance and disappearance of glucose (Ra, Rd), endogenous glucose production (EGP), oxidative and non-oxidative glucose disposal, carbohydrate and lipid oxidation, energy expenditure.

SECONDARY OUTCOMES:
muscle mitochondrial oxidative capacity (in vivo and ex vivo) | 30 days after supplementation
  In vivo: Phosphocreatine levels will be measured by P-MRS (before, during, and after exercise) as a marker for in vivo mitochondrial function in the vastus lateralis muscle.
  Ex vivo mitochondrial function in skeletal muscle will be measured by oxygen consumption in muscle fibres (muscle biopsy) on lipid-derived and carbohydrate-derived substrates.
intramyocellular lipid content | 30 days after supplementation
  Skeletal muscle lipid accumulation measured by immunohistochemistry in muscle biopsy from vastus lateralis muscle
intrahepatic lipid content | 30 days after supplementation
  Intrahepatic lipid content measured with H-MRS
intracardiac lipid content | 30 days after supplementation
  Intracardiac lipid content measured with H-MRS
heart function | 30 days after supplementation
  Cardiac function: diastolic and systolic heart function will be measured with ultrasound
brown adipose tissue activity | 34 days after supplementation
  subjects will be exposed to an individualized cooling protocol, after which an 18F-FDG PET/CT scan is made

OTHER OUTCOMES:
Maximal aerobic capacity (VO2max) | 27 days after supplementation
Blood pressure | 30 days after supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Ligt M, Bruls YMH, Hansen J, Habets MF, Havekes B, Nascimento EBM, Moonen-Kornips E, Schaart G, Schrauwen-Hinderling VB, van Marken Lichtenbelt W, Schrauwen P. Resveratrol improves ex vivo mitochondrial function but does not affect insulin sensitivity or brown adipose tissue in first degree relatives of patients with type 2 diabetes. Mol Metab. 2018 Jun;12:39-47. doi: 10.1016/j.molmet.2018.04.004. Epub 2018 Apr 18. PMID 29706321